CLINICAL TRIAL: NCT00436722
Title: Study of ATEGE-Fresenius Induction in Liver Transplantation Followed by Tacrolimus Weaning.
Brief Title: Induction Treatment Followed by Immunosuppression Withdrawal in Liver Transplantation: A Comparative Trial
Acronym: ATEGE-LIVER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Experimental arm (induction + low dose tacrolimus) not effective.
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fresenius AG (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Miguel navasa, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2005-005635-10
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Liver Diseases
Keywords: Liver; Transplantation; Tolerance; Induction; Tacrolimus; Liver transplantation; Adult
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ATG (Fresenius Biotech) — ATG-Fresenius 9 mg/kg at induction
  Other Names: ATeGe; Anti-lymphocyte immunoglobulin

SUMMARY:
This is a randomized, controlled trial in liver transplantation in which conventional immunosuppressive treatment will be compared with a therapeutic strategy consisting in pre-transplant antibody-mediated T cell depletion followed by reduced calcineurin inhibitor usage. The working hypothesis is that antibody induction followed by calcineurin inhibitor minimization may promote development of tolerogenic mechanisms allowing the eventual withdrawal of all immunosuppressive therapy.

DETAILED DESCRIPTION:
This is an open-label randomised controlled study in which patients will be randomised according to a 1:1 ratio to receive conventional immunosuppressive treatment or induction treatment plus reduced tacrolimus dosage. All transplanted patients enrolled in the study will be followed during 12 months and evaluated according to an intention-to-treat approach.

* Specific Aim 1: To determine the proportion of liver recipients in whom tacrolimus usage can be significantly reduced 1 year after transplantation. Patients will be considered as successfully receiving a reduced tacrolimus regimen if this drug is given as a single dose every other day, or at the most administered as a single dose daily with trough levels < 5ng/mL.
* Specific Aim 2: To determine the effect of induction treatment plus minimized immunosuppression on graft and patient survival.
* Specific Aim 3: To determine the impact of induction treatment plus minimized immunosuppression on the development of: acute and chronic allograft rejection, hepatitis C virus graft recurrence, opportunistic infections, bone fractures, kidney failure, tacrolimus-related neurotoxicity, dyslipidemia and arterial hypertension.
* Specific Aim 4: To establish whether the use of ATG induction followed by reduced doses of tacrolimus differentially affects anti-donor immune responses and/or promotes the development of T cell dependent immunoregulatory networks.
* Conventional immunosuppressive protocol:

  1. Methylprednisolone iv 500 mg before laparotomy, and 500 mg at the time of reperfusion.
  2. Methylprednisolone iv according to the following schedule: postoperative day 1 200 mg, day 2 160mg, day 3 120 mg, day 4 80 mg, day 5 40 mg, and thereafter 20 mg oral prednisone.
  3. Oral tacrolimus q12h starting on postoperative day 1 in order to reach trough drug levels between 10 and 15 ng/mL. These levels will be maintained in this range during the first month after transplantation. Subsequently, tacrolimus levels will be gradually reduced as follows: : month 1-3: 8-15 ng/ml; month 4-12: 7-12 ng/ml; afterwards: 5-10 ng/ml.
  4. Progressive prednisone withdrawal between month 6 and 9 after transplantation.
  5. Treatment of acute rejection episodes: according to our conventional clinical protocol. All efforts must be done in order to histologically document the rejection episode. Hence, empirical treatment should be avoided if possible.
* Induction protocol:

  1. ATG-Fresenius 9mg/kg pre-transplantation, preceded by administration of 500 mg iv methylprednisolone. Infusion of ATG-F will be started whenever the surgeon confirms the suitability of the graft, and will take place during 6 hours.
  2. Oral tacrolimus q12h, starting on postoperative day 1 at the required dosages in order to reach through drug levels between 5 and 12 ng/mL
  3. Reduction of tacrolimus dosages starting 3 months after transplantation in stable patients with no evidences of graft rejection in the previous 60 days, and according to the following protocol:

     * posttransplant month 3: 1 dose per day
     * posttransplant month 6: 1 dose every 48 hours
     * posttransplant month 9: ½ dose every 48 hours
     * posttransplant month 12: evaluate the possibility of complete drug withdrawal or alternatively establish the optimal maintenance dose.
  4. Treatment of acute rejection episodes: mild to moderate acute rejection episodes: re-start 1-2 daily doses of tacrolimus. Severe acute rejection episodes or those mild to moderate episodes that do not improve after 10 days of treatment: 1-2 daily doses of tacrolimus plus methylprednisolone 0.5-1 g for 3 days. Resolution of the rejection episode will be followed by resumption of the above mentioned protocol. If a new rejection episode takes place, after treatment of the acute episode no further attempts to reduce tacrolimus dosages will be attempted. In all cases rejection will be confirmed by liver biopsy.
  5. Patients suffering from hepatitis C virus infection will be treated as above, unless alpha-interferon treatment is considered. In this case, daily tacrolimus will be administered.
  6. All patients will receive CMV prophylaxis with iv ganciclovir for 14 days and oral valganciclovir to complete 3 months after transplantation.
* Sample collection during the study period

In addition to routine diagnostic tests, all enrolled patients will undergo the following procedures:

* Cryopreservation of donor spleen cells to measure anti-donor immune responses.
* HCV viral load quantification pre-transplantation and at post-transplant months 1, 6 and 12.
* All patients will undergo liver biopsy 1 year after transplantation and yearly thereafter. In addition, HCV positive patients will be undergo liver biopsy 3 months after transplantation. A portion of all liver biopsies will be cryopreserved for gene expression studies.
* Anti-donor and anti-HCV T cell immune responses will be quantified before transplantation, and 6 and 12 months after transplantation by gamma-interferon ELISpot assay.
* Peripheral blood mononuclear cells will be harvested and cryopreserved before transplantation, 6 months and 12 months after transplantation to perform gene expression and flow cytometry studies.
* A sample of recipient DNA will be cryopreserved to perform DNA polymorphism studies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Recipient of a primary liver graft
* Absence of any of our exclusion criteria

Exclusion Criteria:

* Pretransplant renal failure, defined as serum creatinine > 1.5 mg/dL
* Severe pretransplant thrombopenia, defined as platelets < 50000/mL
* Combined liver-kidney transplantation
* Autoimmune hepatitis, primary biliary cirrhosis or primary sclerosing cholangitis as causes of liver transplantation
* Chronic hepatic encephalopathy
* Living donor liver transplantation
* Recipient with human immunodeficiency virus infection
* Severe pretransplant leukopenia, defined as < 1500 leukocytes/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who can significantly decrease the doses of tacrolimus 1 year after transplantation (as defined by: tacrolimus administered on alternate days, or daily with trough levels below 5 ng/mL. | 1 year

SECONDARY OUTCOMES:
Graft survival | 1 year
Patient survival | 1 year
Incidence of opportunistic infections | 1 year
Incidence of acute/chronic rejection | 1 year
Incidence of hypertension, renal failure, diabetes, hyperlipidemia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sanchez-Fueyo, Principal Investigator — Hospital Clinic Barcelona, Barcelona, Spain
Locations (1):
- Hospital Clinic Barcelona, University of Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Benitez CE, Puig-Pey I, Lopez M, Martinez-Llordella M, Lozano JJ, Bohne F, Londono MC, Garcia-Valdecasas JC, Bruguera M, Navasa M, Rimola A, Sanchez-Fueyo A. ATG-Fresenius treatment and low-dose tacrolimus: results of a randomized controlled trial in liver transplantation. Am J Transplant. 2010 Oct;10(10):2296-304. doi: 10.1111/j.1600-6143.2010.03164.x. PMID 20883560